CLINICAL TRIAL: NCT04864106
Title: Comprehensive Preoperative Airway Grading
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Michael Froelich, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-300004915; UAB (Other: Anesthesiology)
Record Dates: First submitted 2020-11-05; First posted 2021-04-28 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Anesthesia Intubation Complication
Keywords: Airway Grading
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Intervention Model Description: We are adding a direct laryngoscopy based airway examination to the routine patient examination. Investigators will have two (complementary) methods of a preoperative airway examination; (a) the traditional Malampati airway examination and (b) the new laryngoscopy based examination. Both airway examination methods will be correlated with the airway grading during the induction of anesthesia (Cormack airway grading). The correlation strength of these two preoperative airway assessment methods and the intraoperative Cormack airway grading will be compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Group (Experimental): Participants will undergo a endoscopic airway assessment in addition to the airway classification using the Mallampati score.
  Interventions: Device: Endoscopic Examination

INTERVENTIONS:
Device: Endoscopic Examination — Endoscopic airway grading using a rigid 75-degree angle laryngoscope.

SUMMARY:
Purpose of study: To contrast and compare the Mallampatti test to a comprehensive airway grading test using a rigid 75-degree angle laryngoscope (CPAG) Study Hypothesis: The investigators hypothesize that the CPAG will have greater sensitivity and specificity for predicting difficulty laryngoscopy as compared to the Mallampati test.

The investigators plan to test this hypothesis by comparing the correlation of (a) airway Mallampati airway grading (predicted airway difficulty) versus (b) CPAG view grading and Cormack Laryngoscopy assessment (observed airway difficulty).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate a comprehensive preoperative airway examination using a 75-degree rigid laryngoscope. (It is important to note that this laryngoscope is routinely used in the speech pathology clinic where patients are not required to provide a written consent because of the limited and non-invasive nature of the examination) The investigators plan to accomplish this by grading a person's airway using a laryngoscopy view and obtain pictures to describe a person's supraglottic airway. The investigators will use these measures to assist the anesthesiologists of the day of surgery with the approach of securing the airway (traditional laryngoscopy versus video-assisted laryngoscopy versus fiberoptic-guided laryngoscopy).

The traditional test and parameters for the assessment of the airway are: The Mallampatti test, the Wilson airway assessment, evaluation of the atlantooccipital joint extension (neck mobility), the thyro-mental distance, the sterno-mental distance, mandibulo-hyoid distance, inter-incisor distance (mouth opening). Other investigators have proposed the use of radiographic assessment methods. These traditional tests are limited by the inability to visualize the posterior pharynx, tongue base, and glottis. Difficulty in intubation can be classified according to the view obtained during direct laryngoscopy into 4 grades. These four grades of laryngoscopic views were defined by Cormack and Lehane. At the present time, no single airway test can provide a high index of sensitivity and specificity for the prediction of a difficult airway. Therefore, it is common practice to use a combination of multiple tests and accept that there is still ambiguity when predicting airway challenges and the best approach to securing an airway.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* 18+
* ASA status 1-4

Exclusion Criteria:

* <18
* patients unwilling to do the comprehensive airway examination
* patients unable to do the comprehensive airway examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-11-06 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Participants comparison of grading scores on the traditional procedure verses the comprehensive airway grading | Preoperatively
  Cormack-Lehane system- Grading I-IV looking at the Vocal Cords and Epiglottis (1 is less restricted visibility, 4 is most restricted visibility)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Froelich, MD, MS, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Shanna Graves, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
To be determined.